CLINICAL TRIAL: NCT03849833
Title: Acute Effect of Vitamin D3 Supplementation on Serum 25(OH)D
Brief Title: Acute Effect of Vitamin D3 Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pameli Datta, Medical Doctor, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Dsupplement2019
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
Keywords: Vitamin D; 25(OH)D; vitamin D3 supplementation; pigment genes
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This is a single-centre, open and non-blinded clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin D3 supplementation (Other): All participants will be selected for treatment with cholecalciferol, vitamin D3 supplementation and included in this single arm
  Interventions: Dietary Supplement: cholecalciferol, Vitamin D3

INTERVENTIONS:
Dietary Supplement: cholecalciferol, Vitamin D3 — Vitamin D3 as dietary supplement

SUMMARY:
The investigators have previously completed a clinical trial with long-term vitamin D3 supplementation in healthy humans during a season with negligible ultraviolet B radiation (UVB) in terms of serum 25-hydroxy vitamin D (25(OH)D) increase. In this study (submitted, unpublished), a temporary increase was identified during the first three weeks. Individually, this temporary increase was found in 14 out of 19 participants. This phenomenon has not been described elsewhere in the literature. This could be possible due to less frequent sampling.

The investigators hypothesized that this phenomenon is actual and not an artefact.

The aim of this study was to investigate the serum 25(OH)D increase after short-term vitamin D3 supplementation in a new group of healthy participants with more frequent 25(OH)D sampling. Furthermore, to investigate the influence of sex, age, weight, height, body mass index (BMI), number of fatty fish meals per week, 25(OH)D start level and 30 genetic parameters.

This is a single-centre, open and non-blinded clinical trial. No randomisation was used, as all participants received identical treatment. 25(OH)D sampling was increased from once a week to twice a week. Demographic data (gender, age, weight, height) was collected/measured and registered in prior to study start. The number of daily consumed fatty fish meals was recorded in a questionnaire.

DETAILED DESCRIPTION:
Background The investigators have previously completed a clinical trial with long-term vitamin D3 supplementation in healthy humans during a season with negligible UVB in terms of serum 25-hydroxy vitamin D (25(OH)D) increase. In this study (submitted, unpublished), a temporary increase was identified during the first three weeks. Individually, this temporary increase was found in 14 out of 19 participants. This phenomenon has not been described elsewhere in the literature. This could be possible due to less frequent sampling.

Study hypothesis The investigators hypothesized that this phenomenon is actual and not an artefact. As this phenomenon was not present in all participants, the investigators also hypothesized that influential parameters could include sex, age, weight, height, body mass index (BMI), number of fatty fish meals per week, 25(OH)D start level and genetic parameters (30 pigment single nucleotide polymorphisms (SNP)).

Study design This is a single-centre, open and non-blinded clinical trial.

Intervention Participants will receive packages containing sufficient vitamin D3 tablets (Cholecalciferol, Apovit, Takeda Pharma A/S, Roskilde, Denmark) to cover the consumption corresponding to one week. They will be instructed to consume one vitamin D3 tablet per day corresponding to 85 microgram (ug) (3400 international unit (IU)).

Methodological aspects

Prior intake of vitamin D supplementation Participant will be instructed to not use vitamin D supplementation or participate in a sun holiday at least three weeks prior to study start and during the study.

Compliance Tablets will be counted each week, where the participant will be given supplementation for the following week to control for compliance and adverse events registered. Participants will be instructed to correct deviations in intake of study medication in between each blood sample period with ± ½ tablet per day. A failure to comply with study medication with more that three tablets per week will lead to exclusion.

Blood analysis Serum 25(OH)D will be analysed on a liquid chromatography tandem mass spectrometer (LC-MS/MS), which is the current most accurate method for this analysis. This method has been cross checked against another clinical laboratory and proven reliable. Serum 25(OH)D will also be analysed by the in-house laboratory for comparison.

Analytical variability To minimize analysis variance, at least triplet analyses (technical replicates) will be performed of 25(OH)D analysis. All 25(OH)D samples from the same subject will be analysed in one batch. An internal standard solution with 25(OH)D will be used in each run.

The total relative standard deviation (SD) varies between 4.9% at 20 nmol/l and 14.1% at 222 nmol/l reflecting experimental variability.

Biological variability By including 7 measuring time points for serum 25(OH)D per participant, the intra-individual variability will be reduced. Serum 25(OH)D is known to variate with season and solar exposure. This study was therefore conducted during winter half-year, when ambient UVB radiation and solar-exposed body areas are negligible at this time of the year (17).

Genetic parameters SNP genotyping. A total of 30 pigment SNPs will be investigated. A subgroup of these SNPs have previously been shown to influence the vitamin D3 supplementation induced 25(OH)D increase (paper submitted, unpublished).

All SNPs were genotyped using the iPLEX1 Gold kit (Agena Bioscience Inc., Germany) as previously described. SNPs with genotype subgroups containing less than five subjects were merged with other allele-sharing subgroups (e.g. genotype AA with AG and not with GG). Heterozygote subgroups with less than five subjects was merged with an allele-sharing subgroup displaying insignificant (P > 0.05) difference in influence on the 25(OH)D increase rate. SNPs with no allele dose effect or dominant allele effect on 25(OH)D were excluded. For SNPs with dominant allele effect, subgroups with no significant differences in influence on 25(OH)D increase rate were merged according to allele sharing.

Selection of participants: eligibility criteria All participants must reside in Denmark.

Statistical considerations

Randomization No randomisation will be used, as the aim of this study is to reproduce a biological phenomenon. Blinding will therefore not be used.

Size of study According to a previous vitamin D3 supplementation study (submitted, unpublished) the difference in 25(OH)D from study start to study end was 48 nanomol per liter (nmol l-1) with an SD of 29 nmol l-1. In this present shorter study with vitamin D3 supplementation, the detectable difference in 25(OH)D was expected to be half of that, i.e. 24 nmol l-1. Given a significance level of 5% and a power of 80 %, 13 participants are required. The investigators aim to include 19 participants, allowing six drop-outs.

Sample size calculation was performed using the program Power and Sample Size Calculation version 3.1.2.2014 available online on the website: http://biostat.mc.vanderbilt.edu/wiki/Main/PowerSampleSize

Data collection All participants will be assigned with a unique study number prior to study start. Demographic data (gender, age, weight and height will be collected/measured and registered prior to study start. The number of daily consumed fatty fish meals was recorded in a questionnaire. All forms will be marked with the participants unique study number. 25(OH)D samples will be analysed after study end. The participant study number linked to participant contact details were held in a separate sheet kept securely and in line with the regulation of the Danish Data Protection Agency.

Background diet and change in diet during intervention The number of daily consumed fatty fish meals was recorded in a questionnaire during the study period as this parameter potentially can influence the primary outcome measure, 25(OH)D increase over time. The questionnaire will be examined for errors to ensure compliance.

Background health status and lifestyle, and changes in health status and lifestyle during intervention The health status of the participants and start of new medication was monitored weekly throughout the study.

Adverse events Mild temporary side effects will not lead to discontinuation of study medication. Participants will be monitored with blood samples measuring ionised calcium and alkaline phosphatase. Adverse events such as hypercalcemia or kidney stone will lead to exclusion from the study.

Statistical analysis Individual data will be tested with the Kolmogorov-Smirnov test to assess whether the data are normally distributed. Normally distributed data will be tested by Student's t-test. Pair-wise comparison of ionised calcium (Ca2+) levels at different time points will be performed using Wilcoxon Signed Ranks test.

The following models will be investigated separately: linear, inverse, quadratic, cubic, power, sigmoid and exponential. Determination of the best suitable model (power model) will be based on R2 values and the accordance between the individual investigations and group investigation of the 25(OH)D increase over time.

Initially, the influence of parameters on the 25(OH)D slope will examined separately. The influence of separate significant parameters is not independent and therefore subsequently investigated by a stepwise forward selection of separate significant parameters deployed in a combined general linear model (GLM) according to P-value.25 The influence of parameters on the occurrence of a temporary peak in the serum 25(OH)D over time will also be investigated.

Data will be statistically analysed using SPSS 24.0 for Windows (SPSS Inc., Chicago, IL, U.S.A.). P < 0.05 will be considered significant. No interim analysis will be performed.

Discussion and interpretation The discussion and interpretation of study results will include a consideration of the important study limitations that constitute a bias and discussion of limitations of generalisation of results.

Conclusions The Conclusion section will be related directly to the initial statement of hypothesis and justified by the accompanying data.

Roles and responsibilities of the research team The authors' responsibilities will be specified as follows: 1) designed the research; 2) conducted the research; 3) analysed and interpreted the data; 4) prepared the manuscript; 5) had primary responsibility for the final content and 6) read and approved the final manuscript. All authors will be requested to report conflicts of interest related to this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* resident in Denmark

Exclusion Criteria:

* any supplementary vitamin D intake within three weeks prior to study start
* use of other supplementary vitamin D than given during the study period;
* sun holiday south of latitude 45 degree North less than three weeks prior to or during the study period;
* use of solarium less than three weeks prior to or during the study period;
* chronic disease;
* skin disease;
* intake of cholesterol-lowering medication;
* pregnancy;
* drug addiction;
* psychiatric disorder;
* physical disabilities;
* serious adverse events such as hypercalcaemia and nephrolithiasis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum 25(OH)D | 3 weeks
  Serum 25(OH)D is a marker of vitamin D increase induced by vitamin D3 supplementation
Model of increase in serum 25(OH)D | 3 weeks
  Model fit of the increase in serum 25(OH)D

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Wulf, Professor, Principal Investigator — Department of Dermatology, D92, Bispebjerg Hospital, 2400 Copenhagen NV, Denmark
Locations (1):
- Department of Dermatology, D92, Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No
Indidividual participant data will be shared if requested at publication.